CLINICAL TRIAL: NCT02497508
Title: A Single Arm Phase II Study of Nivolumab in Patients With Recurrent Malignant Pleural Mesothelioma: Interim Biopsy Analysis to Determine Efficacy. Acronym: NivoMes Study
Brief Title: Nivolumab in Patients With Recurrent Malignant Mesothelioma
Acronym: NivoMes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N14MPN
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: progressive disease after at least 1 course of chemotherapy
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab (Experimental): Nivolumab will be administered 2 weekly by intravenous infusion in a dose of 3 mg/kg
  Interventions: Drug: nivolumab

INTERVENTIONS:
Drug: nivolumab
  Other Names: BMS-936558

SUMMARY:
This is a prospective, single arm, phase II trial in previously treated patients with MPM who are considered candidates for immunotherapy and repeat thoracoscopies/transthoracic biopsies. Nivolumab will be administered 3 mg/kg q2 weeks by intravenous injection.

The administration of nivolumab as monotherapy will improve DCR form 20% to 40% at 12 weeks when compared to DCR of patients treated with best supportive care based on historical controls.

DETAILED DESCRIPTION:
Patients will undergo pre- and post-treatment thoracoscopies/biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological diagnosed malignant pleural mesothelioma and age >18 years.
* Progressive disease after at least one course of chemotherapy.
* Previous chemotherapy or experimental therapy ≥ 4 weeks ago.
* Medically suitable for limited surgical intervention (pleural biopsies up to limited pleurectomy).
* Not considered candidates for trimodality treatment (as part of a study).
* Measurable or evaluable disease (see tumor response assessment).
* Ability to understand the study and give signed informed consent prior to beginning of protocol specific procedures including the approval of a second thoracoscopy or transthoracic pleural biopsy after the third course.
* Radiotherapy is allowed when this is given for palliation, the interval is > 12 weeks and not all tumor is within the irradiation field.
* WHO performance status 0 or 1 (see appendix 1).
* Adequate organ function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

  * Hematology: Neutrophil count >= 1.5 x 109/l, Platelets >= 150 x 109/l, Hemoglobin >= 6,0 mmol/l.
  * Chemistry: Total serum bilirubin ≤ 1.5 times within the upper limits of normal (ULN); ASAT and ALAT <= 2.5x ULN, AP (alkaline phosphatases) < 5x ULN (unless bone metastases are present in the absence of any liver disease).

Age and Reproductive Status

* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception to avoid pregnancy during treatment and for 23 weeks after the last dose of investigational drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the first dose of nivolumab.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year during treatment and for a period of 31 weeks after the last dose of investigational drug.
* Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception.

Exclusion Criteria:

* Active uncontrolled infection, severe cardiac dysfunction or uncorrectable bleeding tendency.
* Inability to perform biopsies of the pleural lesions.
* Symptomatic peripheral neuropathy >= grade 2 according to NCI CTC, version 4.0.
* Presence of symptomatic CNS metastases.
* Unstable peptic ulcer, unstable diabetes mellitus or other serious disabling condition.
* Impaired renal function: creatinine clearance less than 50ml/min.
* Concomitant administration to any other experimental drugs under investigation.
* Patients are excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients are excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immuno-suppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients are excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
DCR | at 12 weeks
  The number of patients that have CR or PR plus the number of patients that have SD, as a percentage of the total number of patients in the study.

SECONDARY OUTCOMES:
PFS | Until progression, every 6 weeks up to 24 weeks.
  The time from the date of start of treatment to the date of the first documented tumor progression as determined by modified RECIST, or death due to any cause.
OS | every 8 weeks until death
  The time from date of start of treatment to the date of death
TTP | Until progression, every 6 weeks up to 24 weeks.
  The time from the date of start of treatment to the time of disease progression.
ORR | Every 6 weeks up to 24 weeks.
  The number of subjects whose best confirmed objective response is a CR or PR, divided by the number of treated subjects.
Safety and tolerability (The incidence of (serious) adverse events) | Participants will be followed fot the duration of the trial, an expected average of 6 weeks
  The incidence of (serious) adverse events
DCR | At 6 months
  The number of patients that have CR or PR plus the number of patients that have SD, as a percentage of the total number of patients in the study.

OTHER OUTCOMES:
Exploratory | At screening and after cycle 3 (day 35-50)
  The effects of nivolumab on tissue samples with respect to influx of immuno-modulating cells and the PD-L1 status of tumors and other possible biomarkers and explore correlations between biomarkers and anti-tumor activity.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Baas, MD, PhD, Principal Investigator — The Netherlands Cancer Institute; Josine Quispel-Janssen, MD, Principal Investigator — The Netherlands Cancer Institute

REFERENCES:
- [Derived] Desai AP, Kosari F, Disselhorst M, Yin J, Agahi A, Peikert T, Udell J, Johnson SH, Smadbeck J, Murphy S, Karagouga G, McCune A, Schaefer-Klein J, Borad MJ, Cheville J, Vasmatzis G, Baas P, Mansfield A. Dynamics and survival associations of T cell receptor clusters in patients with pleural mesothelioma treated with immunotherapy. J Immunother Cancer. 2023 Jun;11(6):e006035. doi: 10.1136/jitc-2022-006035. PMID 37279993